CLINICAL TRIAL: NCT00493025
Title: Phase II Study in Operable Adenocarcinoma of the Esophagus to Measure Response Rate and Toxicity of Preoperative Combined Modality Paclitaxel (Taxol®, Bristol-Myers Squibb), Cisplatin (Platinol®, Abbott Laboratories), ZD1839 (IRESSA®) and Radiotherapy Followed by Postoperative ZD1839
Brief Title: Paclitaxel, Cisplatin, Gefitinib, and Radiation Therapy Followed by Surgery and Gefitinib in Treating Patients With Locally Advanced Cancer of the Esophagus or Gastroesophageal Junction That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to early stopping rule-Low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0386; P30CA006973 (NIH); JHOC-J0386; 04-02-20-03 (Other: JHM IRB); ZENECA-IRUSIRES0304; CDR0000549896 (Other: other)
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Gefitinib; Paclitaxel; Chemotherapy, Adjuvant; Radiotherapy

ARMS (1):
- Paclitaxel, Cisplatin, ZD1839 and Radiotherapy (Experimental): Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  Interventions: Drug: cisplatin; Drug: gefitinib; Drug: paclitaxel; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — Cisplatin IV
Drug: gefitinib — Gefitinib IV
  Other Names: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
Drug: paclitaxel — Paclitaxel IV
  Other Names: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
Procedure: adjuvant therapy — Postoperative ZD1839
  Other Names: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
Radiation: radiation therapy — Radiotherapy
  Other Names: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving these treatments before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving gefitinib after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving paclitaxel, cisplatin, gefitinib, and radiation therapy followed by surgery and gefitinib works in treating patients with locally advanced cancer of the esophagus or gastroesophageal junction that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pathologic complete response rate in patients with resectable, locally advanced adenocarcinoma of the esophagus or gastroesophageal junction treated with neoadjuvant paclitaxel, cisplatin, gefitinib, and radiotherapy followed by surgery and adjuvant gefitinib.

Secondary

* Determine the survival of patients treated with this regimen.
* Determine the safety and tolerability of this regimen in these patients.
* Determine time to disease progression in patients treated with this regimen.
* Determine the plasma pharmacokinetics of unbound gefitinib in these patients.
* Conduct exploratory studies to determine if EGFR pathway component expression and activation correlates with response to therapy and survival of these patients.
* Determine if treatment with gefitinib alters the EGFR pathway in these patients.

OUTLINE: This is a prospective study.

* Neoadjuvant therapy: Patients receive oral gefitinib beginning 14 days prior to the start of chemoradiotherapy and continuing until 7 days prior to surgery (10-12 weeks). Patients also receive paclitaxel IV over 1 hour and cisplatin IV over 2-3 hours on days 1, 8, 15, 22, and 29. Patients also undergo radiotherapy 5 days a week for 5 weeks.
* Surgery: Patients undergo surgical resection 4-6 weeks after the completion of neoadjuvant therapy.
* Adjuvant therapy: Patients receive gefitinib once a day beginning 2-8 weeks after surgery and continuing for up to 1 year in the absence of disease progression or unacceptable toxicity.

Blood samples are obtained at baseline and periodically during study for pharmacokinetic studies. Tumor tissue samples are obtained by core biopsy at baseline for biomarker correlative studies. Samples are analyzed by IHC to measure expression and activation of EGFR-signaling pathway biomarkers in pretreatment esophageal tumor tissue, including EGFR and phosphorylated (p)-EGFR, ERK and p-ERK, Akt and p-Akt, p70s6k and p-p70s6k, and p27.

After completion of study therapy, patients are followed periodically for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the esophagus or gastroesophageal junction meeting the following criteria:

  * Newly diagnosed disease
  * Surgically resectable tumor
  * Primary esophageal tumor < 20 cm below the incisors
  * Tumor extending ≤ 2 cm into the cardia
* Stage T2-3, N0-1, M0-1a tumor, as determined by imaging studies and biopsy

  * Documentation by endoscopic ultrasound, endoscopy, and CT scan of the chest and abdomen required
  * Any lesion suspicious for metastasis must be biopsied
  * M1a disease (i.e., celiac nodal metastasis) is allowed if other eligibility criteria are met
  * T4 disease (i.e., involvement of the pleura, pericardium, or diaphragm) allowed provided it is considered resectable
* No CNS metastasis
* ECOG performance status 0-1
* Granulocyte count > 1,000/mm³
* Platelet count > 75,000/mm³
* Creatinine clearance > 60 mL/min
* Total bilirubin < 1.5 mg/dL
* No concurrent illness likely to preclude protocol therapy or surgical resection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy Exclusion Criteria
* Known severe hypersensitivity to gefitinib or any of its excipients
* Evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* Evidence of other significant clinical disorder or laboratory finding that would preclude study participation
* Evidence of clinically active interstitial lung disease
* Chronic, stable radiographic changes that are asymptomatic are eligible
* Prior or concurrent malignancy except basal cell or squamous cell skin cancer, cervical cancer, or any other curatively treated malignancy from which the patient has been disease-free and has a survival prognosis of > 5 years
* Preexisting peripheral neuropathy > grade 1
* Incomplete healing from prior oncologic or other major surgery
* Prior chemotherapy, radiotherapy, or surgery for this cancer
* More than 30 days since prior nonapproved or investigational drugs
* Concurrent phenytoin, carbamazepine, barbiturates, rifampin, phenobarbital, or Hypericum perforatum (St. John's wort)
* Concurrent oral retinoids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene A. Forastiere, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel, Cisplatin, ZD1839 and Radiotherapy: Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  cisplatin: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  gefitinib: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Posto ZD1839
  paclitaxel: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  gene expression analysis: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  immunohistochemistry staining method: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  laboratory biomarker analysis: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  pharmacological study: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  adjuvant therapy: Combined Modality Paclitaxel, Cisplatin,
Period: Overall Study
Arm/Group | Paclitaxel, Cisplatin, ZD1839 and Radiotherapy
Started | 19
Completed | 0 (Trial stopped due to early stopping rule)
Not Completed | 19
Not completed — Physician Decision | 19

BASELINE CHARACTERISTICS:
Groups:
- Paclitaxel, Cisplatin, ZD1839 and Radiotherapy: Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  cisplatin: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  gefitinib: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  paclitaxel: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  gene expression analysis: Combined Modality Paclitaxel, Cisplatin, ZD1839 Radiotherapy Followed by Postoperative ZD1839
  immunohistochemistry staining method: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  laboratory biomarker analysis: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  pharmacological study: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  adjuvant therapy: Combined Modality Paclitaxel, Cisplatin,
Arm/Group | Paclitaxel, Cisplatin, ZD1839 and Radiotherapy
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] — Trial stopped due to early stopping rule, no data analysis completed.
  years | 67 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate to the Neoadjuvant Regimen
Description: Study closed due to early stopping rule. Patient data was not analyzed. No additional information is available to report
Time Frame: 5 years
Population: Study terminated due to early stopping rule. Therefore, data was not collected to assess this outcome measure
Groups:
- Paclitaxel, Cisplatin, ZD1839 and Radiotherapy: Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  cisplatin: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  gefitinib: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  paclitaxel: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  gene expression analysis: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  immunohistochemistry staining method: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  laboratory biomarker analysis: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  pharmacological study: Combined Modality Paclitaxel, Cisplatin, ZD1839 and Radiotherapy Followed by Postoperative ZD1839
  adj therapy: Combined Modality Paclitaxel, Cisplatin,
Arm/Group | Paclitaxel, Cisplatin, ZD1839 and Radiotherapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Toxicity as Assessed by NCI CTC v2.0
Time Frame: 5 years
Population: Study terminated due to early stopping rule. Therefore, data was not collected to assess this outcome measure
Arm/Group | Paclitaxel, Cisplatin, ZD1839 and Radiotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Safety and Tolerability of This Regimen
Time Frame: 5 years
Population: Study terminated due to early stopping rule. Therefore, data was not collected to assess this outcome measure
Arm/Group | Paclitaxel, Cisplatin, ZD1839 and Radiotherapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Progression
Time Frame: 5 years
Population: Study terminated due to early stopping rule. Therefore, data was not collected to assess this outcome measure
Arm/Group | Paclitaxel, Cisplatin, ZD1839 and Radiotherapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Survival
Time Frame: 5 years
Population: Study terminated due to early stopping rule. Therefore, data was not collected to assess this outcome measure
Arm/Group | Paclitaxel, Cisplatin, ZD1839 and Radiotherapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Correlation Between EGFR Pathway Component Expression and Activation With Pathologic Complete Response and Survival
Time Frame: 5 years
Population: Study terminated due to early stopping rule. Therefore, data was not collected to assess this outcome measure
Arm/Group | Paclitaxel, Cisplatin, ZD1839 and Radiotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Paclitaxel, Cisplatin, ZD1839 and Radiotherapy
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
Study was closed due to early stopping rule.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes